CLINICAL TRIAL: NCT04916899
Title: Study to Evaluate the Safety of the Use of doTBal (Rifampicin, Isoniazid, Pyrazinamide and Ethambutol) in Patients With Tuberculosis: Conduction of an Intensive Pharmacovigilance Program
Brief Title: Safety of doTBal® in Patients With Tuberculosis: Conduction of an Intensive Pharmacovigilance Program
Status: Completed | Type: Observational
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: DoTBal_FVI_001
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB; Tuberculosis treatment; adverse events; pharmacovigilance
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Isoniazid; Pyrazinamide; Ethambutol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Rifampicin/ Isoniazid/ Pyrazinamide/ Ethambutol: Pharmaceutical Form: Tablets Dosage: 150 mg / 75 mg / 400 mg / 300 mg Administration way: oral
  Interventions: Drug: Rifampicin/ Isoniazid/ Pyrazinamide/ Ethambutol

INTERVENTIONS:
Drug: Rifampicin/ Isoniazid/ Pyrazinamide/ Ethambutol — Form: Tablets Dosage: 150 mg / 75 mg / 400 mg / 300 mg Adminstration way: Oral
  Other Names: doTbal®

SUMMARY:
Phase IV, observational, cohort, prospective study. With duration according to the indicated scheme, 6 months of treatment (2 intensive months and 4 months of sotén) for pulmonary tuberculosis. Follow-up with patients will continue for a month after completion of the indicated scheme.

DETAILED DESCRIPTION:
The objective of the study was to detect and analyze the adverse events presented during the administration of the drug doTBal® in patients of the Health Centers of the Ministry of Health of the municipalities of Colima, Tecomán and Manzanillo, of the State of Colima. All patients detected in the selected centers that are indicated treatment with doTBal® under the TAES (Strictly Supervised Shortened Treatment) regimen or who are already on this drug (according to their clinical record), will be asked to participate in the study explaining to them the same and requesting their informed consent in writing. In the case of minors, they will also be asked to provide their informed assent.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with a diagnosis of active pulmonary tuberculosis.
* Over 12 years old.
* Patients who are being treated with doTBal® under the TAES (Strictly Supervised Shorter Treatment) regimen.
* Informed consent (and in the case of minors informed consent) signed.

Exclusion Criteria:

* Withdrawal of informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients over 12 years old, who are being trated with doTBal® under strictly supervised shorter treatment regimen and sign informes consent.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To detect adverse events | 23 months
  To detect the adverse events presented during the administration of the drug doTBal®
Frequency of occurrence of adverse events | 23 months
  Determine the frequency of appearance of each adverse event detected with the administration of the drug doTBal®
Severity of each of the adverse events | 23 months
  Determine the severity of each of the adverse events during the administration of the drug doTBal®
Causality of each of the adverse events | 23 months
  Analyze the causality of each of the adverse events detected during the administration of the drug doTBal® (using the Tree-orange algorithm)
Apparatus and systems affected with adverse events | 23 months
  Analyze the apparatus and systems affected with adverse events during drug administration of doTBal®
Factors associated with the presentation of adverse events | 23 months
  Analyze other factors associated with the presentation of adverse events during doTBal® administration, such as age, sex, pregnancy, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Maldonado Hernández, MS., Principal Investigator — Centro de Salud Colima; Martha Castrejón, M.D, Principal Investigator — Centro de Salud Tecomán; José G Maya Campos, M.D, Principal Investigator — Centro Avanzado de Atención Primaria a la Salud; Adara M Cárdenas Sánchez, M.D, Principal Investigator — Centro de Salud Urbano Salangua
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumberg HM, Burman WJ, Chaisson RE, Daley CL, Etkind SC, Friedman LN, Fujiwara P, Grzemska M, Hopewell PC, Iseman MD, Jasmer RM, Koppaka V, Menzies RI, O'Brien RJ, Reves RR, Reichman LB, Simone PM, Starke JR, Vernon AA; American Thoracic Society, Centers for Disease Control and Prevention and the Infectious Diseases Society. American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America: treatment of tuberculosis. Am J Respir Crit Care Med. 2003 Feb 15;167(4):603-62. doi: 10.1164/rccm.167.4.603. No abstract available. PMID 12588714
- See also: NOM-220-SSA1-2016: 2.1.11 — https://www.dof.gob.mx/nota_detalle.php?codigo=5601541&fecha=30/09/2020
- See also: Buenas Prácticas de Farmacovigilancia para las Américas, 2008 — https://www3.paho.org/hq/index.php?option=com_docman&view=download&category_slug=documentos-8499&alias=33513-buenas-pra-cticas-farmacovigilancia-ame-ricas-2010-513&Itemid=270&lang=es
- See also: NORMA Oficial Mexicana NOM-006-SSA2-2013, Para la prevención y control de la tuberculosis. — http://dof.gob.mx/nota_detalle.php?codigo=5321934&fecha=13/11/2013